CLINICAL TRIAL: NCT03068325
Title: Trauma-Focused Equine-Assisted Therapy (TF-EAT) for Veterans With PTSD
Acronym: TF-EAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Research Foundation for Mental Hygiene, Inc. (Other)
Collaborators: Columbia University (Other)
Responsible Party: Principal Investigator, Yuval Y Neria, Professor of Medical Psychology, Research Foundation for Mental Hygiene, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB # 7232
Record Dates: First submitted 2017-02-26; First posted 2017-03-01 (Actual); Results first posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Posttraumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

ARMS (1):
- EAT-PTSD (Experimental): Manualized Equine-Assisted Treatment for PTSD (EAT-PTSD) seeks to increase affective awareness of self and others, improve communication, help regulate emotional response, improve critical thinking/problem solving, and increase self-confidence/self-efficacy while engaging with the horses.
  Interventions: Other: EAT-PTSD

INTERVENTIONS:
Other: EAT-PTSD

SUMMARY:
This study seeks to examine feasibility, acceptability, safety, and preliminary efficacy of Equine-Assisted Therapy for veterans with posttraumatic stress disorder (EAT-PTSD). While several well-studied, validated treatments for PTSD exist, some individuals find these treatments ill-suited, ineffective, or undesirable. EAT is an alternative therapy widely used by organizations, such as PATH International Equine Services, that endorse its effectiveness for treating a variety of mental health issues. These claims have drawn criticism because the published research contains glaring methodological flaws, making it difficult to assess how effective these therapies actually are (Anestis et al., 2014). Equine-assisted therapies present a unique treatment modality that might effectively treat PTSD, particularly for individuals who have difficulty with other treatment modalities. In EAT, a psychotherapist and equine specialist work together to help the patients negotiate interactions with a horse using structured interventions or activities.

DETAILED DESCRIPTION:
In this pilot study the investigators will develop the EAT intervention and determine whether research methods (evaluation interviews, assessment measures, videotaping procedures) are acceptable to participants. Specifically, the investigators will focus on issues such as session length, appropriateness of the "content" for treatment of PTSD, ordering of session content, adherence to the manual of the equine therapeutic team (based on observations made during supervision and feedback from the consultants), and will detail logistics of data collection and how best to record the sessions (camera angles, etc.).

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 70
* Current DSM-5 diagnosis of PTSD as determined by a) full criteria met on CAPS, and b) clinical assessment
* Able to give consent, fluent in English

Exclusion Criteria:

* History of psychiatric diagnosis of psychotic disorder, unstable bipolar disorder
* Elevated depression of clinical concern and/or score of >25 on the Hamilton Rating Scale for Depression
* At elevated risk for suicide based on history and current mental state
* History of substance/alcohol use disorder at severe level within the past six months, and current diagnosis of substance/alcohol use disorder at a moderate level within past two months
* Fear of horses or other large animals
* Orthopedic or other physical conditions and/or limitations that prevent people from walking unassisted and/or walking freely in the ring.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2019-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yuval Neria, PhD, Principal Investigator — Columbia University Irving Medical Center, New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

REFERENCES:
- [Derived] Fisher PW, Lazarov A, Lowell A, Arnon S, Turner JB, Bergman M, Ryba M, Such S, Marohasy C, Zhu X, Suarez-Jimenez B, Markowitz JC, Neria Y. Equine-Assisted Therapy for Posttraumatic Stress Disorder Among Military Veterans: An Open Trial. J Clin Psychiatry. 2021 Aug 31;82(5):21m14005. doi: 10.4088/JCP.21m14005. PMID 34464523
- [Derived] Zhu X, Suarez-Jimenez B, Zilcha-Mano S, Lazarov A, Arnon S, Lowell AL, Bergman M, Ryba M, Hamilton AJ, Hamilton JF, Turner JB, Markowitz JC, Fisher PW, Neria Y. Neural changes following equine-assisted therapy for posttraumatic stress disorder: A longitudinal multimodal imaging study. Hum Brain Mapp. 2021 Apr 15;42(6):1930-1939. doi: 10.1002/hbm.25360. Epub 2021 Feb 5. PMID 33547694
- [Derived] Arnon S, Fisher PW, Pickover A, Lowell A, Turner JB, Hilburn A, Jacob-McVey J, Malajian BE, Farber DG, Hamilton JF, Hamilton A, Markowitz JC, Neria Y. Equine-Assisted Therapy for Veterans with PTSD: Manual Development and Preliminary Findings. Mil Med. 2020 Jun 8;185(5-6):e557-e564. doi: 10.1093/milmed/usz444. PMID 32034416

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Ninety-seven individuals were assessed for eligibility in the study, but 34 were excluded as a result of not meeting study inclusion criteria, leaving 63 participants to proceed into study enrollment.
Groups:
- EAT-PTSD: Manualized EAT-PTSD seeks to increase affective awareness of self and others, improve communication, help regulate emotional response, improve critical thinking/problem solving, and increase self-confidence/self-efficacy while engaging with the horses.
Period: Overall Study
Arm/Group | EAT-PTSD
Started | 63
Completed | 58
Not Completed | 5
Not completed — Lost to Follow-up | 5

BASELINE CHARACTERISTICS:
Arm/Group | EAT-PTSD
Number analyzed (Participants) | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.01 (12.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 40
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 16
  Black/African-American | 26
  Other | 15
  Prefer not to respond | 6
Index Trauma [Count of Participants; unit: Participants]
  Combat-related | 27
  Military sexual trauma | 23
  Physical assault | 9
  Sexual assault | 1
  Child abuse | 23
  Traumatic accident | 4
  Natural disaster | 1
  Traumatic sudden loss | 7
  Other | 16
Service Era [Count of Participants; unit: Participants]
  1960-1969 | 6
  1970-1979 | 14
  1980-1989 | 20
  1990-1999 | 20
  2000-2009 | 31
  2010-2019 | 15
Military Conflicts [Count of Participants; unit: Participants]
  Vietnam/Korea | 10
  OEF/OIF | 23
  Other | 5
  None | 25

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Clinician-Administered PTSD Scale at 8 Weeks
Description: Change in symptoms of PTSD as assessed by the Clinician-Administered PTSD Scale for DSM-5 (CAPS-5, severity rating ranging from 0-80 with higher scores indicating more severe PTSD) in a clinical interview
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | EAT-PTSD
Number analyzed (Participants) | 63
score on a scale
  Baseline | 38.6 (8.1)
  8 weeks | 26.9 (12.4)

ADVERSE EVENTS:
Time Frame: Study period (baseline to 3-month follow-up; total: five months)
Arm/Group | EAT-PTSD
All-Cause Mortality (participants affected / at risk) | 0/63
Serious Adverse Events (participants affected / at risk) | 0/63
Other Adverse Events (participants affected / at risk) | 0/63

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-09): https://cdn.clinicaltrials.gov/large-docs/25/NCT03068325/Prot_SAP_000.pdf